CLINICAL TRIAL: NCT04538560
Title: Preimplantation Genetic Testing for Aneuploidy by Next-generation Sequencing of Polar Bodies in Advanced Maternal Age With Poor Ovarian Responders: a Randomized Clinical Trial (Preliminary Experiments)
Brief Title: Preimplantation Genetic Testing for Aneuploidy of Polar Bodies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P2020002
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Subfertility
Keywords: poor ovarian respond，; advanced age; Preimplantation Genetic Testing
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polar body biopsy group (Experimental): The study group will undergo polar body biopsy, and the NGS technology will be used to evaluate the polar body euploidy and then predict the euploidy of the oocyte. Embryo transfer priority according to the NGS test results and morphological scores.
  Interventions: Procedure: polar body biopsy
- Control group (No Intervention): The control group will undergo routine culture and the transfer priority is determined according to the morphological score only.

INTERVENTIONS:
Procedure: polar body biopsy — Undergo polar body biopsy, and the NGS technology will be used to evaluate the polar body euploidy and then predict the euploidy of the oocyte. Embryo transfer priority according to the NGS test results and morphological scores.
  Arms: Polar body biopsy group

SUMMARY:
This study intends to randomly group the patients with advanced maternal age and poor ovarian response, and the study group will undergo polar body biopsy, and the next-generation sequencing(NGS) technology will be used to evaluate the polar body euploidy and then predict the euploidy of the oocyte. Embryo transfer priority according to the NGS test results and morphological scores. In the control group undergo routine culture and the transfer priority is determined according to the morphological score only. The transfer of frozen embryos at the cleavage or blastocyst stage was permitted. Cumulative live birth rate, miscarriage rate and time required to obtain a live birth up to two ovulatory cycles in a year.

ELIGIBILITY:
Inclusion Criteria:

* patients between their 36th and 42st birthdays;
* absence of any type of genetic abnormality in the patient's personal and family history;
* MⅡ oocytes: 2-9 .

Exclusion Criteria:

* treatment involving donor oocytes;
* any type of genetic abnormality or family history of genetic abnormality in subject or partner;
* with assisted reproductive technology and pregnancy contraindications and with diseases that have a definite effect on pregnancy;
* poor embryo quality in previous cycles;
* Preimplantation genetic testing for aneuploidy(PGT-A) cycles;
* MⅡ oocytes ≥10 or ≤ 1;
* three or more previous failed IVF or Intracytoplasmic sperm injection(ICSI) cycles.

Ages: 36 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative live birth rate | 22 months

SECONDARY OUTCOMES:
abortion rate | 22 months
time required to obtained a live birth | 22 months

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive and Genetic Hospital of Citic-xiangya, Changsha, Hunan, China